CLINICAL TRIAL: NCT02796963
Title: Institute for Global Health & Infectious Diseases (IGHID) 11604 - Crowdsourcing to Promote HIV Testing: A Stepped Wedge Randomized Controlled Trial to Evaluate Promoting HIV Testing in China
Brief Title: Crowdsourcing A Public Health Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); UNC-South China STD Research Training Center (Unknown); UNC Center for AIDS Research (Unknown); SESH Global (Unknown); Guangdong Provincial Center for Skin Diseases and STI Control (Unknown); London School of Hygiene and Tropical Medicine (Other); University of Bristol (Other); Shandong University (Other); Shandong Province Centers for Disease Control and Prevention (Other); Guangdong Center for Disease Prevention and Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-0851; R01AI114310 (NIH)
Record Dates: First submitted 2016-05-23; First posted 2016-06-13 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-02

CONDITIONS: HIV
Keywords: HIV; MSM; test uptake; crowdsourcing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Intervention (Experimental): Men will be exposed immediately to a comprehensive intervention promoting HIV testing.
  Interventions: Behavioral: Crowdsourced intervention
- Delayed Intervention (Experimental): Men will be exposed to a comprehensive intervention promoting HIV testing after a delay period.
  Interventions: Behavioral: Crowdsourced intervention; Behavioral: Traditional intervention campaign

INTERVENTIONS:
Behavioral: Crowdsourced intervention — The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
Behavioral: Traditional intervention campaign — The pre-intervention period will include conventional HIV testing campaigns organized by local CDC, Community-Based Organization (CBO), and partners. These are typically designed by experts and social marketing companies.
  Other Names: Conventional HIV testing campaign
  Arms: Delayed Intervention

SUMMARY:
The purpose of this stepped wedge randomized controlled trial is to evaluate the effectiveness of a crowdsourced intervention on promoting HIV testing among young Chinese men who have sex with men (MSM). The crowdsourced intervention will include an open contest, judging to determine finalists and prizes, a designathon, and contest-based MSM engagement. The hypothesis is that a crowdsourced intervention will be superior to conventional HIV test uptake campaigns in eliciting HIV test uptake.

DETAILED DESCRIPTION:
This study will use an adaptation of the stepped wedge randomized controlled trial design. A total of eight major metropolitan cities will implement the crowdsourced intervention. These cities will be chosen based on the following criteria: 1) previous Centers for Disease Control and Prevention (CDC) MSM sentinel surveillance site; 2) capacity for campaign implementation; 3) capacity for intervention implementation at the community level. Four cities will implement more intensive in-person events to promote engagement (Guangzhou, Shenzhen in Guangdong Province, Qingdao, and Jinan in Shandong Province) during survey intervention stage. The Randomized controlled trial (RCT) will be evaluated using two different sources of data: 1) online survey data from MSM in the eight cities prior to and after the intervention; 2) CDC routine surveillance data in the eight cities prior to and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Currently living and planning to live in one of the eight cities used in the study in the next 12 months.
* Not living with HIV
* No HIV test in the past three months
* Born biologically male and identify as either male or transgender female
* Had anal or oral sex with men at least once during their lifetime
* 16 years or older
* Willing to provide cell phone number
* Complete the informed consent document

Exclusion Criteria:

* Women are excluded from this study

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1381 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tucker, MD, PhD, Principal Investigator — jdtucker@med.unc.edu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tang W, Han L, Best J, Zhang Y, Mollan K, Kim J, Liu F, Hudgens M, Bayus B, Terris-Prestholt F, Galler S, Yang L, Peeling R, Volberding P, Ma B, Xu H, Yang B, Huang S, Fenton K, Wei C, Tucker JD. Crowdsourcing HIV Test Promotion Videos: A Noninferiority Randomized Controlled Trial in China. Clin Infect Dis. 2016 Jun 1;62(11):1436-1442. doi: 10.1093/cid/ciw171. Epub 2016 Apr 29. PMID 27129465
- [Background] Zhang Y, Kim JA, Liu F, Tso LS, Tang W, Wei C, Bayus BL, Tucker JD. Creative Contributory Contests to Spur Innovation in Sexual Health: 2 Cases and a Guide for Implementation. Sex Transm Dis. 2015 Nov;42(11):625-8. doi: 10.1097/OLQ.0000000000000349. PMID 26462186
- [Derived] Ong JJ, Booton RD, Tucker JD, Tang W, Vickerman P, Zhang L, Mitchell KM. Economic evaluation of improving HIV self-testing among MSM in China using a crowdsourced intervention: a cost-effectiveness analysis. AIDS. 2023 Mar 15;37(4):671-678. doi: 10.1097/QAD.0000000000003457. Epub 2022 Dec 9. PMID 36729711
- [Derived] Tang W, Wei C, Cao B, Wu D, Li KT, Lu H, Ma W, Kang D, Li H, Liao M, Mollan KR, Hudgens MG, Liu C, Huang W, Liu A, Zhang Y, Smith MK, Mitchell KM, Ong JJ, Fu H, Vickerman P, Yang L, Wang C, Zheng H, Yang B, Tucker JD. Crowdsourcing to expand HIV testing among men who have sex with men in China: A closed cohort stepped wedge cluster randomized controlled trial. PLoS Med. 2018 Aug 28;15(8):e1002645. doi: 10.1371/journal.pmed.1002645. eCollection 2018 Aug. PMID 30153265
- [Derived] SESH Study Group; Tucker JD. Crowdsourcing to promote HIV testing among MSM in China: study protocol for a stepped wedge randomized controlled trial. Trials. 2017 Oct 2;18(1):447. doi: 10.1186/s13063-017-2183-1. PMID 28969702
- See also: University of North Carolina website — http://www.unc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 28, 2016, and followed until August 21, 2017. A total of 1,381 participants were enrolled. Of these, 203, 139, 134 and 203 were recruited from Guangzhou, Jiangmen, Zhuhai and Shenzhen, respectively, while 180, 189, 182 and 151 were recruited from Yantai, Jinan, Qingdao and Jining, respectively.
Pre-assignment Details: Overall, the survey link was clicked 36,863 times from 25,141 independent Internet Protocol (IP) addresses, and a total of 2,112 eligible participants finished the questionnaire (many people clicked the survey link but withdrew before the eligible screening). Among these 2,112 participants, 1381 were eligible for the study.
Units Other Than Participants: City
Groups:
- Immediate Intervention: Based on the pre-determined randomization schedule, 383 participants from Guangzhou and Yantai were assigned to the first intervention group to receive a crowdsourced intervention in months 1-3.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
- Delayed Intervention 1: Based on the pre-determined randomization schedule, 328 participants from Jiangmen and Jinan were assigned to the delayed intervention group 2 to receive a crowdsourced intervention in months 4-6.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
- Delayed Intervention 2: Based on the pre-determined randomization schedule, 316 participants from Zhuhai and Qingdao were assigned to the delayed intervention group 2 to receive a crowdsourced intervention in months 7-9.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
- Delayed Intervention 3: Based on the pre-determined randomization schedule, 354 participants from Shenzhen and Jining were assigned to delayed intervention group 3 to receive a crowdsourced intervention in months 10-12.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
Period: Overall Study
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Started | 383; 2 City | 328; 2 City | 316; 2 City | 354; 2 City
First Follow up | 293; 2 City | 279; 2 City | 257; 2 City | 291; 2 City
Second Follow up | 280; 2 City | 260; 2 City | 255; 2 City | 293; 2 City
Third Follow up | 276; 2 City | 237; 2 City | 245; 2 City | 286; 2 City
Fourth Follow up | 275; 2 City | 233; 2 City | 236; 2 City | 263; 2 City
HIV Sero Converted | 19; 2 City | 19; 2 City | 11; 2 City | 19; 2 City
Completed | 294; 2 City | 252; 2 City | 247; 2 City | 282; 2 City
Not Completed | 89; 0 City | 76; 0 City | 69; 0 City | 72; 0 City
Not completed — Lost to Follow-up | 89 | 76 | 69 | 72

BASELINE CHARACTERISTICS:
Groups:
- Immediate Intervention: Guangzhou and Yantai city. Intervention in months 1-3: A crowdsourcing contest to solicit optimal images/concepts/taglines; a designathon to formulate optimal HIV testing campaigns; a process of localization unique to each of the eight cities.
- Delayed Intervention 1: Jiangmen and Jinan city. Intervention in months 4-6: A crowdsourcing contest to solicit optimal images/concepts/taglines; a designathon to formulate optimal HIV testing campaigns; a process of localization unique to each of the eight cities.
- Delayed Intervention 2: Zhuhai and Qingdao city. Intervention in months 7-9: A crowdsourcing contest to solicit optimal images/concepts/taglines; a designathon to formulate optimal HIV testing campaigns; a process of localization unique to each of the eight cities.
- Delayed Intervention 3: Shenzhen and Jining city. Intervention in months 10-12: A crowdsourcing contest to solicit optimal images/concepts/taglines; a designathon to formulate optimal HIV testing campaigns; a process of localization unique to each of the eight cities.
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3 | Total
Number analyzed (Participants) | 383 | 328 | 316 | 354 | 1381
Age, Customized [Count of Participants; unit: Participants]
  16-20 years | 65 | 78 | 81 | 87 | 311
  21-25 years | 146 | 118 | 94 | 111 | 469
  26-30 years | 100 | 80 | 80 | 95 | 355
  >30 years | 72 | 52 | 61 | 61 | 246
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 364 | 314 | 301 | 334 | 1313
  Transgender individuals | 19 | 14 | 15 | 20 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 383 | 328 | 316 | 354 | 1381
Region of Enrollment [Count of Participants; unit: Participants]
  China | 383 | 328 | 316 | 354 | 1381
Marital Status [Count of Participants; unit: Participants]
  Never married | 337 | 290 | 268 | 299 | 1194
  Married | 46 | 38 | 48 | 55 | 187
Annual income, US$ [Count of Participants; unit: Participants]
  <3000 | 75 | 82 | 64 | 64 | 285
  3000-6000 | 75 | 86 | 71 | 67 | 299
  6001-9500 | 133 | 88 | 93 | 120 | 434
  9501-12500 | 65 | 50 | 52 | 67 | 234
  >12500 | 35 | 22 | 36 | 36 | 129
Highest education [Count of Participants; unit: Participants]
  High school or below | 132 | 106 | 118 | 127 | 483
  College or beyond | 251 | 222 | 198 | 227 | 898
Sexual orientation [Count of Participants; unit: Participants]
  Gay | 296 | 225 | 230 | 229 | 980
  Bisexual | 87 | 103 | 86 | 125 | 401
Disclosure of sexual orientation [Count of Participants; unit: Participants]
  Disclosed to others | 262 | 205 | 209 | 222 | 898
  Not disclosed to others | 121 | 123 | 107 | 132 | 483
Condomless sex [Count of Participants; unit: Participants] — Ever had condomless sex in the past three months
  Participants
    No | 101 | 92 | 85 | 98 | 376
    Yes | 282 | 236 | 231 | 256 | 1005
Syphilis testing [Count of Participants; unit: Participants] — Had syphilis test in the past three months
  Participants
    No | 360 | 317 | 301 | 335 | 1313
    Yes | 23 | 11 | 15 | 19 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Men Who Have Sex With Men (MSM) Reporting HIV Testing in the Past Three Months
Description: This will be assessed by self-report during a follow-up survey
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 56 | 85 | 122 | 128

2. Secondary Outcome: Number of Men Reporting Condomless Sex at 3 Months Post-intervention
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 74 | 52 | 62 | 60

3. Secondary Outcome: HIV Testing Social Norms
Description: HIV testing social norms will be measured using six survey items that are each on a five-point Likert scale. Increased HIV testing social norms will be defined as having an increase from baseline in any two of these six survey items and dichotomized accordingly. Number of men who report higher score of social norms when comparing their pre-intervention and post-intervention values
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 214 | 181 | 175 | 190

4. Secondary Outcome: Change in HIV Testing Self-efficacy
Description: Number of men who report higher levels of self-efficacy when comparing their pre-intervention and post-intervention HIV testing norms
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 200 | 173 | 153 | 181

5. Secondary Outcome: Community Engagement/ MSM Community Affiliation
Description: Number of men, defined as an increase in closer affiliation with the MSM community (i.e., tongzhi circle, gay online networks or groups) when comparing their pre-intervention and post-intervention periods.
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 190 | 148 | 157 | 176

6. Secondary Outcome: Number of Men Reporting Engaged in HIV Testing Community Campaign in the Past 3 Months
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 269 | 246 | 226 | 236

7. Secondary Outcome: Number of Men Reporting Being Self-tested for HIV in the Last 3 Months Post-intervention
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 32 | 68 | 94 | 107

8. Secondary Outcome: Mean Score of Anticipated HIV Stigma
Description: Measured by a 7-item version of the anticipated HIV stigma scale, designed to measure the extent to which participants anticipated negative intrapersonal and interpersonal consequences were they to contract HIV in the future. All seven items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate greater anticipated stigma.
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Scores on a scale | 2.06 (0.65) | 2.06 (0.70) | 2.11 (0.66) | 2.08 (0.69)

9. Secondary Outcome: Number of Men Reporting Being Tested for Syphilis in the Last 3 Months Post-intervention
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 22 | 29 | 37 | 50

10. Secondary Outcome: Number of Men Reporting Using Weibo in the Past Three Months Post-intervention to Give or Receive Information About HIV Testing
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 49 | 56 | 44 | 46

11. Secondary Outcome: Number of Men Reporting Using Wechat in the Past Three Months Post-intervention to Give or Receive Information About HIV Testing
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 117 | 101 | 97 | 102

12. Secondary Outcome: Number of Men Reporting Using Tencent QQ (QQ) in the Past Three Months Post-intervention to Give or Receive Information About HIV Testing
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 47 | 71 | 44 | 49

13. Secondary Outcome: Number of Men Reporting Using Mobile Apps in the Past Three Months Post-intervention to Give or Receive Information About HIV Testing
Description: Frequency of men, defined as the number of men who reported using mobile apps in the past three months to give or receive information about HIV testing comparing their pre-intervention and post-intervention engagement
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 71 | 54 | 63 | 81

14. Secondary Outcome: Number of Men Reporting Received HIV Self-testing Kits in the Last 3 Months Post-intervention
Time Frame: From implementation roll-out to three months after implementation of crowdsourced intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
Number analyzed (Participants) | 293 | 260 | 245 | 263
Participants | 91 | 73 | 89 | 120

ADVERSE EVENTS:
Time Frame: 1 year (July 28, 2016- August 20, 2017)
Groups:
- Immediate Intervention: Based on the pre-determined randomization schedule, 383 participants from Guangzhou and Yantai were assigned to the first intervention group to receive a crowdsourced intervention in months 1-3.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
  No adverse outcome was reported.
- Delayed Intervention 1: Based on the pre-determined randomization schedule, 328 participants from Jiangmen and Jinan were assigned to the delayed intervention group 2 to receive a crowdsourced intervention in months 4-6.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
  No adverse outcome was reported.
- Delayed Intervention 2: Based on the pre-determined randomization schedule, 316 participants from Zhuhai and Qingdao were assigned to the delayed intervention group 2 to receive a crowdsourced intervention in months 7-9.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
  No adverse outcome was reported.
- Delayed Intervention 3: Based on the pre-determined randomization schedule, 354 participants from Shenzhen and Jining were assigned to delayed intervention group 3 to receive a crowdsourced intervention in months 10-12.
  Crowdsourced intervention: The crowdsourced intervention is composed of three phases that cumulatively draw on crowd wisdom to engage the community: (1) a crowdsourcing contest to solicit optimal images/concepts/taglines; (2) a designathon to formulate optimal HIV testing campaigns; (3) a process of localization unique to each of the eight cities.
  No adverse outcome was reported.
Arm/Group | Immediate Intervention | Delayed Intervention 1 | Delayed Intervention 2 | Delayed Intervention 3
All-Cause Mortality (participants affected / at risk) | 0/383 | 0/328 | 0/316 | 0/354
Serious Adverse Events (participants affected / at risk) | 0/383 | 0/328 | 0/316 | 0/354
Other Adverse Events (participants affected / at risk) | 0/383 | 0/328 | 0/316 | 0/354

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02796963/Prot_SAP_000.pdf